CLINICAL TRIAL: NCT01896531
Title: A Randomized, Phase II, Placebo-controlled Study of Ipatasertib (GDC-0068), an Inhibitor to Akt, in Combination With Fluoropyrimidine Plus Oxaliplatin in Patients With Locally Advanced or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: A Study of Ipatasertib (GDC-0068) in Combination With Fluoropyrimidine Plus Oxaliplatin in Participants With Advanced or Metastatic Gastric or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO28341; 2012-002080-10 (EudraCT Number)
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Results first posted 2022-02-17 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Fluorouracil; ipatasertib; Leucovorin; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ipatasertib + mFOLFOX6 (Experimental): Participants will receive oral ipatasertib on Days 1 to 7 of each 14-day cycle in combination with mFOLFOX6, administered on Day 1 of each cycle.
  Interventions: Drug: 5-Fluorouracil; Drug: Ipatasertib; Drug: Leucovorin; Drug: Oxaliplatin
- Placebo + mFOLFOX6 (Placebo Comparator): Participants will receive the placebo equivalent to ipatasertib on Days 1 to 7 of each 14-day cycle in combination with mFOLFOX6, administered on Day 1 of each cycle.
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Placebo

INTERVENTIONS:
Drug: 5-Fluorouracil — Participants will receive bolus and infusional 5-fluorouracil on Day 1 of each 14-day cycle (as a part of mFOLFOX6 therapy), until disease progression or unacceptable toxicity. The infusion times for infusional 5-fluorouracil may be determined per local and/or institutional standards and product labeling.
Drug: Ipatasertib — Participants will receive ipatasertib, 600 milligrams (mg) orally once daily on Days 1 to 7 of each 14-day cycle until disease progression or unacceptable toxicity.
  Arms: Ipatasertib + mFOLFOX6
Drug: Leucovorin — Participants will receive leucovorin or equivalent substitute orally, on Day 1 of each 14-day cycle (as a part of mFOLFOX6 therapy), until disease progression or unacceptable toxicity.
Drug: Oxaliplatin — Participants will receive oxaliplatin via intravenous (IV) infusion on Day 1 of each 14-day cycle (part of mFOLFOX6 therapy). Oxaliplatin will be discontinued after completion of 8 cycles
Drug: Placebo — Participants will receive matching oral placebo capsules once daily on Days 1 to 7 of each 14-day cycle until disease progression or unacceptable toxicity.
  Arms: Placebo + mFOLFOX6

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled study will evaluate the efficacy of ipatasertib in combination with oxaliplatin, 5-fluorouracil, and leucovorin (modified FOLFOX6 [mFOLFOX6]) chemotherapy in participants with advanced or metastatic gastric or gastroesophageal junction (GEJ) cancer. Participants will be randomized to receive either ipatasertib or placebo orally daily on Days 1 to 7 of each 14-day cycle in combination with mFOLFOX6 on Day 1 of each cycle.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically documented, inoperable locally advanced or metastatic or recurrent gastric/GEJ adenocarcinoma, not amenable to curative therapy
* Measurable disease, according to RECIST v1.1
* Life expectancy greater than or equal to (>/=) 12 weeks
* Adequate hematologic and organ function

Exclusion Criteria:

* Previous chemotherapy for inoperable locally advanced or metastatic gastric/GEJ adenocarcinoma. Participants may have received prior neoadjuvant or adjuvant chemotherapy and/or radiation treatment for locally advanced gastric/GEJ adenocarcinoma, provided all treatments were completed >/= 6 months prior to randomization.
* Known human epidermal growth factor receptor 2 (HER2)-positive gastric/GEJ adenocarcinoma
* Radiation treatment within 28 days of randomization. Participants who have received palliative radiation treatment to peripheral sites (eg, bone metastases) within 28 days of randomization may be enrolled in the study if they have recovered from all acute, reversible effects and with notification of the Medical Monitor.
* Previous therapy for gastric/GEJ adenocarcinoma with Akt, phosphatidylinositol 3-kinase (PI3K), and/or mammalian target of rapamycin (mTOR) inhibitors
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomization or anticipation of need for a major surgical procedure during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2013-08-14 (Actual); Primary Completion 2015-06-03 (Actual); Study Completion 2021-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (34):
- United States (3):
  - Univ of Calif, Los Angeles; Hematology/Oncology, Los Angeles, California
  - Massachusetts General Hospital;Oncology, Boston, Massachusetts
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Institut Gustave Roussy; Departement Oncologie Medicale, Villejuif, France
- Germany (3):
  - Charité-Universitätsm. Berlin; Med. Klinik mit Schwerpunkt Hämatologie, Onkologie und Tumorimmunolo., Berlin
  - Medizinische Hochschule Hannover; Zentrum Innere Medizin; Abt. Hämatologie u. Onkologie, Hanover
  - Universitatsklinik Heidelberg; Universitätshautklinik und Nationales Centrum für Tumorerkrankungen, Heidelberg
- Queen Mary Hospital; Dept. of Clinical Oncology, Hong Kong, Hong Kong
- Italy (3):
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST); Oncologia Medica A, Genoa, Liguria
  - Azienda Ospedaliero Universitaria Pisana; Uff. Sperim. Clin. U.O. Farmaceutica, Pisa, Tuscany
  - IRCCS Istituto Oncologico Veneto (IOV); Oncologia Medica Seconda, Padua, Veneto
- Malaysia (3):
  - Hospital Universiti Sains Malaysia [Neurology], Kubang Kerian, Kelantan
  - Gleneagles Medical Centre, George Town
  - University Malaya Medical Centre; Clinical Oncology Unit,, Kuala Lumpur
- Singapore (2):
  - National Cancer Centre; Medical Oncology, Singapore
  - Oncocare Cancer Centre, Singapore
- South Korea (8):
  - Kyungpook National University Hospital, Daegu
  - Gachon Medical School Gil Medical Centre; Internal Medicine, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center; Medical Oncology, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hosp; Dept Internal Med Hem Onc, Seoul
  - Yonsei Uni College of Medicine, Severance Hospital; Internal Medicine Dept., Seoul
  - St Vincent'S Hospital; Oncology, Suwon
- Spain (3):
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (3):
  - National Cheng Kung Univ Hosp, Tainan
  - National Taiwan Uni Hospital; Dept of Oncology, Taipei
  - Chang Gung Medical Foundation - Linkou; Division of Hematology- Oncology, Taoyuan District
- United Kingdom (4):
  - Royal Marsden Hospital; Dept of Med-Onc, London
  - Sarah Cannon Research Institute, London
  - Mount Vernon Hospital; Centre For Cancer Treatment, Northwood
  - The Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] Bang YJ, Kang YK, Ng M, Chung HC, Wainberg ZA, Gendreau S, Chan WY, Xu N, Maslyar D, Meng R, Chau I, Ajani JA. A phase II, randomised study of mFOLFOX6 with or without the Akt inhibitor ipatasertib in patients with locally advanced or metastatic gastric or gastroesophageal junction cancer. Eur J Cancer. 2019 Feb;108:17-24. doi: 10.1016/j.ejca.2018.11.017. Epub 2018 Dec 25. PMID 30592991

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 33 centers in 11 countries.
Pre-assignment Details: Total 153 participants were randomized in this study, of which 152 participants received treatment.
Groups:
- Ipatasertib + mFOLFOX6: Ipatasertib was administered at a dose of 600 milligrams (mg) orally once daily, beginning on Day 1 of Cycle 1 through Day 7 of each 14-day cycle until the participant experienced disease progression or intolerable toxicity. Following ipatasertib administration on Day 1 of each cycle, the participant then received mFOLFOX6 in the following order: oxaliplatin as an 85 milligram per square-meter (mg/m^2) intravenous (IV) infusion on Day 1 every 14 days with co-administration of leucovorin at 400 mg/m^2 or equivalent substitute. The participant then received 5-fluorouracil (5-FU) as a 400 mg/m^2 bolus infusion followed by 5-FU as a 2400 mg/m^2 continuous IV infusion (or 5-FU as a 1200 mg/m^2/day continuous IV infusion). Following Cycle 8, oxaliplatin was discontinued.
- Placebo + mFOLFOX6: Placebo matched to ipatasertib was administered orally once daily, beginning on Day 1 of Cycle 1 through Day 7 of each 14-day cycle until the participant experienced disease progression or intolerable toxicity. Following placebo administration on Day 1 of each cycle, the participant then received mFOLFOX6 in the following order: oxaliplatin as an 85 mg/m^2 IV infusion on Day 1 every 14 days with co-administration of leucovorin at 400 mg/m^2 or equivalent substitute. The participant then received 5-FU as a 400 mg/m^2 bolus infusion followed by 5-FU as a 2400 mg/m^2 continuous IV infusion (or 5-FU as a 1200 mg/m^2/day continuous IV infusion). Following Cycle 8, oxaliplatin was discontinued.
Period: Overall Study
Arm/Group | Ipatasertib + mFOLFOX6 | Placebo + mFOLFOX6
Started | 71 | 82
Treated | 70 | 82
Completed | 0 | 0
Not Completed | 71 | 82
Not completed — Death | 57 | 59
Not completed — Lost to Follow-up | 3 | 0
Not completed — Non-compliance | 0 | 1
Not completed — Study Ended by Sponsor | 7 | 20
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Death Prior to Treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipatasertib + mFOLFOX6 | Placebo + mFOLFOX6 | Total
Number analyzed (Participants) | 71 | 82 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (11.4) | 61.4 (11.0) | 59.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 41
  Male | 52 | 60 | 112
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 67 | 81 | 148
  Not Stated | 2 | 1 | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 43 | 45 | 88
  White | 25 | 36 | 61
  Other | 2 | 0 | 2
  Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) in All Randomized Participants and Participants With PTEN Loss Tumors at Primary Analysis
Description: PFS was defined as the time from randomization to the first occurrence of disease progression (as determined using RECIST Version 1.1 and assessed by the investigator), or death from any cause on study. Progressive disease (PD): At least a 20% increase in the sum of diameters of target lesions, and the sum must also demonstrate an absolute increase of at least 5 mm or progression of non-target lesions. Death on study was defined as death from any cause within 30 days of the last dose of study treatment regimen. Kaplan-Meier estimates were used for evaluation.
Time Frame: Screening, at the end of Cycle 4 (cycle = 14 days) and every fourth cycle thereafter until disease progression or death, whichever occurred first, assessed up to approximately 1.75 years
Population: The randomized population was defined as all participants who were randomized in the study. Randomized participants with PTEN loss tumors were also analyzed. For the primary analysis, PTEN loss was defined as the condition "Perc Cells Cytoplasmic Stain Int 0" of greater than or equal to 10.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Ipatasertib + mFOLFOX6 | Placebo + mFOLFOX6
Number analyzed (Participants) | 71 | 82
months
  All Randomized Participants | 6.57 [5.72 to 7.52] | 7.52 [6.24 to 8.11]
  Participants With PTEN Loss Tumors: number analyzed (Participants) | 15 | 21
  Participants With PTEN Loss Tumors | 7.10 [5.39 to 9.92] | 7.39 [6.51 to 14.69]
Statistical Analysis 1: Comparison: Ipatasertib + mFOLFOX6 vs Placebo + mFOLFOX6; All randomized participants; Test type: Superiority — Unstratified analysis; p = 0.56, Log Rank; Hazard Ratio (HR) = 1.12, 90% CI 2-sided [0.81 to 1.55]
Statistical Analysis 2: Comparison: Ipatasertib + mFOLFOX6 vs Placebo + mFOLFOX6; Participants with PTEN loss tumors; Test type: Superiority — Unstratified analysis; p = 0.86, Log Rank; Hazard Ratio (HR) = 1.07, 90% CI 2-sided [0.54 to 2.11]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. Kaplan-Meier estimates were used for evaluation.
Time Frame: Baseline up to end of study (up to approximately 7.5 years)
Population: All randomized participants, randomized participants with PTEN loss tumors and randomized participants who were Akt diagnostic-positive (Akt Dx+) were analyzed. For the final analysis, PTEN loss was defined as the condition "Perc Cells Cytoplasmic Stain Int 0" of greater than 10.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Ipatasertib + mFOLFOX6 | Placebo + mFOLFOX6
Number analyzed (Participants) | 71 | 82
months
  Randomized | 11.96 [10.28 to 14.55] | 15.31 [13.54 to 16.92]
  PTEN Loss Tumors: number analyzed (Participants) | 14 | 15
  PTEN Loss Tumors | 14.82 [11.99 to 18.40] | 21.78 [14.13 to NA] — NA: not estimable due to low number of events
  Akt Dx+: number analyzed (Participants) | 23 | 23
  Akt Dx+ | 11.66 [9.92 to 18.40] | 17.22 [12.71 to 23.29]
Statistical Analysis 1: Comparison: Ipatasertib + mFOLFOX6 vs Placebo + mFOLFOX6; All randomized participants; Test type: Superiority — Unstratified analysis; p = 0.0234, Log Rank; Hazard Ratio (HR) = 1.52, 90% CI 2-sided [1.12 to 2.07]
Statistical Analysis 2: Comparison: Ipatasertib + mFOLFOX6 vs Placebo + mFOLFOX6; Participants with PTEN loss tumors; Test type: Superiority — Unstratified analysis; p = 0.2867, Log Rank; Hazard Ratio (HR) = 1.66, 90% CI 2-sided [0.75 to 3.65]
Statistical Analysis 3: Comparison: Ipatasertib + mFOLFOX6 vs Placebo + mFOLFOX6; Participants who are Akt Dx+; Test type: Superiority — Unstratified analysis; p = 0.1369, Log Rank; Hazard Ratio (HR) = 1.66, 90% CI 2-sided [0.94 to 2.93]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate was defined as the percentage of participants achieving either a complete response (CR) or a partial response (PR) based on the investigator assessment using RECIST v 1.1. CR: disappearance of all target lesions and all pathological lymph nodes below 10 mm. Partial response (PR): At least a 30% decrease in the sum of diameters of target lesions.
Time Frame: Screening, at the end of Cycle 4 (cycle = 14 days) and every fourth cycle thereafter until disease progression or death, whichever occurred first, up to end of study (up to approximately 7.5 years)
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Ipatasertib + mFOLFOX6 | Placebo + mFOLFOX6
Number analyzed (Participants) | 71 | 82
percentage of participants
  Randomized | 52.1 [41.74 to 62.35] | 57.3 [48.02 to 66.59]
  PTEN Loss Tumors: number analyzed (Participants) | 14 | 15
  PTEN Loss Tumors | 50.0 [26.36 to 73.64] | 73.3 [50.00 to 87.82]
  Akt Dx+: number analyzed (Participants) | 23 | 23
  Akt Dx+ | 52.2 [33.51 to 70.39] | 56.5 [38.05 to 72.67]
Statistical Analysis 1: Comparison: Ipatasertib + mFOLFOX6 vs Placebo + mFOLFOX6; All randomized participants; Test type: Superiority; p = 0.5202, Cochran-Mantel-Haenszel; Difference in Response Rates = -5.20, 90% CI 2-sided [-18.46 to 8.06]
Statistical Analysis 2: Comparison: Ipatasertib + mFOLFOX6 vs Placebo + mFOLFOX6; Participants with PTEN loss tumors; Test type: Superiority; p = 0.2035, Cochran-Mantel-Haenszel; Difference in Response Rates = -23.33, 90% CI 2-sided [-52.24 to 5.58]
Statistical Analysis 3: Comparison: Ipatasertib + mFOLFOX6 vs Placebo + mFOLFOX6; Participants who are Akt Dx+; Test type: Superiority; p = 0.7697, Cochran-Mantel-Haenszel; Difference in Response Rates = -4.35, 90% CI 2-sided [-28.48 to 19.79]

4. Secondary Outcome: Duration of Objective Tumor Response
Description: Duration of objective tumor response in participants with measurable soft tissue disease at baseline was defined as the time from first observation of an objective tumor response until first observation of disease progression, as assessed by the investigator per modified RECIST Version 1.1. PD: At least a 20% increase in the sum of diameters of target lesions, and the sum must also demonstrate an absolute increase of at least 5 mm or progression of non-target lesions.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Ipatasertib + mFOLFOX6 | Placebo + mFOLFOX6
Number analyzed (Participants) | 37 | 47
months
  Randomized | 4.63 [4.01 to 5.52] | 5.85 [4.47 to 6.90]
  PTEN Loss Tumor: number analyzed (Participants) | 7 | 11
  PTEN Loss Tumor | 4.70 [4.27 to NA] — NA: not estimable due to low number of events | 5.98 [4.86 to 10.94]
  Akt Dx+: number analyzed (Participants) | 12 | 13
  Akt Dx+ | 4.70 [3.84 to 14.78] | 6.80 [4.86 to 10.71]
Statistical Analysis 1: Comparison: Ipatasertib + mFOLFOX6 vs Placebo + mFOLFOX6; All randomized participants; Test type: Superiority — Unstratified analysis; p = 0.5974, Log Rank; Hazard Ratio (HR) = 1.14, 90% CI 2-sided [0.76 to 1.73]
Statistical Analysis 2: Comparison: Ipatasertib + mFOLFOX6 vs Placebo + mFOLFOX6; Participants with PTEN loss tumors; Test type: Superiority — Unstratified analysis; p = 0.5385, Log Rank; Hazard Ratio (HR) = 0.71, 90% CI 2-sided [0.28 to 1.79]
Statistical Analysis 3: Comparison: Ipatasertib + mFOLFOX6 vs Placebo + mFOLFOX6; Participants who are Akt Dx+; Test type: Superiority — Unstratified analysis; p = 0.6097, Log Rank; Hazard Ratio (HR) = 0.78, 90% CI 2-sided [0.35 to 1.75]

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. Death on study was defined as death from any cause within 30 days of the last dose of study treatment regimen.
Time Frame: Baseline until end of study (up to approximately 7.5 years)
Population: The safety population was defined as all randomized participants who received at least one dose of ipatasertib/placebo or mFOLFOX6, with participants grouped according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Ipatasertib + mFOLFOX6 | Placebo + mFOLFOX6
Number analyzed (Participants) | 70 | 82
Participants | 70 | 80

6. Secondary Outcome: Serum Concentration of Ipatasertib
Time Frame: Day 1 at 1 hour and 4 hours post-dose; Day 5, pre-dose and 2 hours post-dose
Population: The pharmacokinetic (PK) population was defined as all participants with evaluable PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ipatasertib + mFOLFOX6
Number analyzed (Participants) | 64
ng/mL
  Day 1: 1 hour post-dose: number analyzed (Participants) | 63
  Day 1: 1 hour post-dose | 506 (550)
  Day 1: 4 hours post-dose | 389 (202)
  Day 5: pre-dose: number analyzed (Participants) | 62
  Day 5: pre-dose | 90.7 (61.0)
  Day 5: 2 hours post-dose: number analyzed (Participants) | 57
  Day 5: 2 hours post-dose | 557 (328)

ADVERSE EVENTS:
Time Frame: Baseline until end of study (up to approximately 7.5 years)
Description: Safety population included treated participants (i.e., participants who received at least one dose of ipatasertib/placebo or mFOLFOX6), with participants allocated to the treatment arm associated with the regimen that they actually received.
Arm/Group | Ipatasertib + mFOLFOX6 | Placebo + mFOLFOX6
All-Cause Mortality (participants affected / at risk) | 57/70 | 59/82
Serious Adverse Events (participants affected / at risk) | 39/70 | 36/82
Other Adverse Events (participants affected / at risk) | 70/70 | 79/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipatasertib + mFOLFOX6 (N=70) | Placebo + mFOLFOX6 (N=82)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0)
ULCERATIVE KERATITIS (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 (4) | 4 (4)
ASCITES (Gastrointestinal disorders) | 0 (0) | 2 (4)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 5 (6) | 3 (3)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 2 (2)
ENTERITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTRIC PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 2 (2) | 1 (1)
ILEUS (Gastrointestinal disorders) | 3 (4) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 1 (1)
INTESTINAL PSEUDO-OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
JEJUNAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 4 (5) | 0 (0)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 2 (3) | 2 (2)
OESOPHAGEAL FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 2 (2)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 0 (0)
VOMITING (Gastrointestinal disorders) | 3 (3) | 4 (5)
ASTHENIA (General disorders) | 1 (1) | 2 (2)
DEATH (General disorders) | 1 (1) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 0 (0)
OBSTRUCTION (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 3 (4) | 3 (3)
BILIARY OBSTRUCTION (Hepatobiliary disorders) | 1 (1) | 0 (0)
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 1 (1) | 0 (0)
APPENDICITIS PERFORATED (Infections and infestations) | 0 (0) | 1 (1)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (1) | 0 (0)
LARGE INTESTINE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1)
PERITONITIS (Infections and infestations) | 0 (0) | 1 (1)
PHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 2 (2)
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1) | 2 (2)
TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CHEMICAL PERITONITIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0)
CACHEXIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 (5) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
HYPERGLYCAEMIC HYPEROSMOLAR NONKETOTIC SYNDROME (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CEREBRAL GAS EMBOLISM (Nervous system disorders) | 0 (0) | 1 (1)
DIABETIC HYPEROSMOLAR COMA (Nervous system disorders) | 1 (1) | 0 (0)
PARAPARESIS (Nervous system disorders) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 2 (2) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY TRACT DISORDER (Renal and urinary disorders) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
VENOUS THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipatasertib + mFOLFOX6 (N=70) | Placebo + mFOLFOX6 (N=82)
ANAEMIA (Blood and lymphatic system disorders) | 14 (27) | 15 (22)
GRANULOCYTOPENIA (Blood and lymphatic system disorders) | 4 (6) | 6 (10)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (4) | 6 (10)
NEUTROPENIA (Blood and lymphatic system disorders) | 21 (38) | 33 (71)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 8 (14) | 11 (22)
VISION BLURRED (Eye disorders) | 2 (2) | 5 (11)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 6 (6) | 3 (5)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 9 (10) | 7 (9)
ABDOMINAL PAIN (Gastrointestinal disorders) | 19 (26) | 20 (34)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 9 (10) | 7 (10)
CONSTIPATION (Gastrointestinal disorders) | 27 (59) | 24 (48)
DIARRHOEA (Gastrointestinal disorders) | 57 (202) | 34 (73)
DRY MOUTH (Gastrointestinal disorders) | 4 (6) | 8 (10)
DYSPEPSIA (Gastrointestinal disorders) | 9 (11) | 17 (22)
DYSPHAGIA (Gastrointestinal disorders) | 7 (13) | 7 (8)
FLATULENCE (Gastrointestinal disorders) | 2 (3) | 5 (6)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 6 (6) | 5 (10)
NAUSEA (Gastrointestinal disorders) | 51 (117) | 51 (133)
STOMATITIS (Gastrointestinal disorders) | 17 (26) | 8 (12)
VOMITING (Gastrointestinal disorders) | 43 (104) | 33 (87)
ASTHENIA (General disorders) | 13 (17) | 16 (27)
CATHETER SITE PAIN (General disorders) | 4 (4) | 5 (7)
CHEST DISCOMFORT (General disorders) | 5 (6) | 2 (3)
CHEST PAIN (General disorders) | 4 (5) | 6 (8)
FATIGUE (General disorders) | 44 (112) | 37 (83)
INFLUENZA LIKE ILLNESS (General disorders) | 4 (4) | 3 (4)
MUCOSAL INFLAMMATION (General disorders) | 13 (46) | 15 (20)
OEDEMA PERIPHERAL (General disorders) | 7 (10) | 8 (13)
PYREXIA (General disorders) | 15 (18) | 9 (10)
TEMPERATURE INTOLERANCE (General disorders) | 7 (8) | 11 (12)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 (10) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 10 (11) | 4 (9)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 7 (9) | 6 (8)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 5 (7) | 10 (15)
BLOOD CREATININE INCREASED (Investigations) | 6 (8) | 4 (6)
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 1 (1) | 5 (8)
GLYCOSYLATED HAEMOGLOBIN INCREASED (Investigations) | 1 (1) | 5 (5)
NEUTROPHIL COUNT DECREASED (Investigations) | 5 (7) | 12 (18)
PLATELET COUNT DECREASED (Investigations) | 6 (10) | 5 (18)
WEIGHT DECREASED (Investigations) | 16 (21) | 9 (13)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 3 (4) | 5 (7)
DECREASED APPETITE (Metabolism and nutrition disorders) | 41 (115) | 41 (92)
DEHYDRATION (Metabolism and nutrition disorders) | 5 (5) | 5 (6)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 14 (23) | 15 (28)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 6 (7) | 5 (7)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 4 (4) | 2 (4)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 11 (14) | 8 (11)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 7 (13) | 4 (7)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 4 (7) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 (9) | 10 (12)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 (14) | 14 (23)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 3 (6) | 7 (8)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (7)
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 (8) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (11)
DIZZINESS (Nervous system disorders) | 15 (18) | 13 (19)
DYSGEUSIA (Nervous system disorders) | 5 (5) | 8 (8)
HEADACHE (Nervous system disorders) | 7 (20) | 8 (16)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 27 (46) | 38 (100)
PARAESTHESIA (Nervous system disorders) | 6 (10) | 6 (6)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 10 (17) | 14 (24)
TASTE DISORDER (Nervous system disorders) | 8 (8) | 7 (7)
ANXIETY (Psychiatric disorders) | 5 (5) | 3 (3)
INSOMNIA (Psychiatric disorders) | 12 (18) | 13 (20)
PROTEINURIA (Renal and urinary disorders) | 5 (7) | 3 (5)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 12 (15)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 10 (16) | 15 (21)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (5)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 5 (6)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (7)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (5)
ALOPECIA (Skin and subcutaneous tissue disorders) | 13 (13) | 20 (22)
DRY SKIN (Skin and subcutaneous tissue disorders) | 5 (7) | 8 (11)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (9)
PRURITUS (Skin and subcutaneous tissue disorders) | 10 (11) | 6 (6)
RASH (Skin and subcutaneous tissue disorders) | 20 (34) | 11 (20)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 4 (6) | 0 (0)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 5 (5)
HYPERTENSION (Vascular disorders) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.